CLINICAL TRIAL: NCT00754637
Title: Microplasty Tibial Tray Multi-Center Data Collection
Brief Title: Microplasty Tibial Tray Data Collection
Acronym: MTT
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn because it no longer fit the business need.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 335
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Joint Disease
Keywords: Joint; Osteoarthritis; Avascular Necrosis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 510(k) Inclusion Criteria: Any person meeting the inclusion criteria for the device may be included in this study. These patients tend to be those seeking relief from painful or debilitating knee joint disease.

SUMMARY:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Microplasty Tibial Tray.

DETAILED DESCRIPTION:
FDA has cleared this device via premarket notification 510(k) K063732. By being CE Marked, the Microplasty Tibial Tray also conforms to the essential requirements of EC Directive 93/42/EEC; in accordance to 13485:2003. The data gathered would be collated and used to provide feedback to design engineers, support marketing efforts, and answer potential questions from reimbursement agencies, and will serve as a part of Biomet's Post Market Surveillance System.

Inclusion/exclusion criteria are identical to those indications and contraindications stated in the FDA approved labeling for the device in 510(k) K063732 Surgical techniques and patient care are to be standard for the surgeon participating in the protocol and should be maintained the same throughout the course of the data-collection. There will be no experimental or investigational devices used. There will be no experimental or investigational surgical techniques used. The devices and products will be used in accordance with their instructions for use and/or approved labeling. Any use of the device or collection of clinical data outside of the United States should comply with all local, state, and/or national and international regulations.

Function will be assessed through the Knee Society Score . Survivorship will be documented by asking the surgeon to document revisions and complications.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be identical to the indications stated in the FDA approved labeling for the device in 510(k) K063732. These indications are stated below:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure.

Patient selection factors to be considered include:

* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions, including control of weight and activity level
* A good nutritional state of the patient, and
* The patient must have reached full skeletal maturity

Non-coated (Interlock®) devices are indicated for cemented application only.

Exclusion Criteria:

The exclusion criteria will be identical to the contraindications stated in the FDA approved labeling for the device in 510(k) K063732. These contraindications are stated below:

Absolute contraindications include: infection, sepsis, and osteomyelitis.

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* Osteoporosis,
* Metabolic disorders which may impair bone formation,
* Osteomalacia,
* Distant foci of infections which may spread to the implant site,
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
* Vascular insufficiency, muscular atrophy, neuromuscular disease,
* Incomplete or deficient soft tissue surrounding the knee.

Biomet Microplasty™ Tibial Trays are contraindicated for use with constrained bearings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of relief frm painful or disabling Joint Disease, and meeting the 510(k) inclusion criteria on the cleared device.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | 5 years

SECONDARY OUTCOMES:
Radiographic Data | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Beres, MD, Study Director — Zimmer Biomet
Locations (1):
- The DeClaire Knee & Orthopaedic Institute, Rochester Hills, Michigan, United States

REFERENCES:
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Amstutz HC, Thomas BJ, Jinnah R, Kim W, Grogan T, Yale C. Treatment of primary osteoarthritis of the hip. A comparison of total joint and surface replacement arthroplasty. J Bone Joint Surg Am. 1984 Feb;66(2):228-41. PMID 6693450
- [Background] Brooks, et al. (Eds.). (2003) The Measurement and Valuation of Health Status Using EQ-5D: A European Perspective. Netherlands: Kluwer Academic Publishers.